CLINICAL TRIAL: NCT05241496
Title: Lidocaine Spray 10% Versus Oral Ibuprofen Tablets in Pain Control During Copper Intrauterine Device Insertion (A Randomized Controlled Trial)
Brief Title: Lidocaine Spray 10% Versus Oral Ibuprofen Tablets in Pain Control During Copper Intrauterine Device Insertion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marina Ramsis Aziz Ghaly (Other)
Responsible Party: Sponsor-Investigator, Marina Ramsis Aziz Ghaly, principal investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AinShams univ
Record Dates: First submitted 2022-01-17; First posted 2022-02-15 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Lidocaine Toxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Marina Ramsis (Experimental): In the other group, 70 women will be randomly assigned for ibuprofen; participants will take 1 tablet (400mg) immediately & clinicians will wait at least 45 minutes before inserting the copper IUD
  Interventions: Diagnostic Test: The spray form may provide easy application and better patient acceptance than other forms of lidocaine administration

INTERVENTIONS:
Diagnostic Test: The spray form may provide easy application and better patient acceptance than other forms of lidocaine administration — Lidocaine in spray form is a simple and convenient local anaesthetic with minimal adverse effects and is often used in dentistry for oral mucosal anaesthesia during minor surgical interventions. The spray form may provide easy application and better patient acceptance than other forms of lidocaine administration. Lidocaine acts by stabilization of the neuronal membrane by inhibiting the ionic fluxes required for the initiation and conduction of impulses, thereby effecting local anesthetic action (Hüseyin Aksoy et al. ,2016 ) .

SUMMARY:
The intrauterine contraceptive device (IUD) is the most commonly used form of reversible contraception worldwide; the predominant type of product, the copper IUD (a plastic T-shaped device with copper affixed to it) was developed over 30 years ago and has become the standard bearer for intrauterine contraception, due to its long-term effectiveness, safety and affordability .

Inconsistent use and discontinuation of contraceptives are major causes of unintended pregnancy . The failure rate of the patch or ring is 20 times higher than that of long acting reversible contraceptives (LARCs) . Increasing acceptability and use of LARC methods like the intrauterine device (IUD) is an important strategy to reduce the risk of unintended pregnancy

DETAILED DESCRIPTION:
The aim of this study is to This study is designed to compare between lidocaine spray 10% and oral ibuprofen as an adequate method for decreasing pain during copper intrauterine contraceptive device insertion .

Research question:

Which of both drugs ( local lidocaine spray 10% or oral ibuprofen tab.) is more effective in decreasing pain during IUD insertion ? Research Hypothesis In this current study, we hypothesize that using of local cervical lidocaine spray 10% prior to IUD insertion will decrease the pain more effectively than ibuprofen tablet 400 mg.

ELIGIBILITY:
Inclusion Criteria:

-Multiparous women in 3rd to 5th day of menstrual cycle 2- Women who were 6 weeks postpartum or if recently pregnant. 3- Accept to participate and provide consent

Exclusion Criteria:

* • A contraindication for IUD use such as a gynecological malignancy , sexually transmitted diseases, pelvic inflammatory disease or undiagnosed abnormal vaginal bleeding.

  * Suspicion of pregnancy .
  * Allergy to lidocaine or ibuprofen .
  * Copper allergy .
  * Any uterine abnormalities distorted uterine cavity as congenital anomalies, endometrial lesions, adenomyosis , and submucous myoma.
  * A psychological or neurological disorder associated with altered pain sensation.
  * MIRENA insertion.
  * Nulliparity.
  * History of failed intrauterine device insertion (uterine perforation, acute expulsion).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 1 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-12-14 (Estimated); Study Completion 2023-10-10 (Estimated)

PRIMARY OUTCOMES:
Self-reported pain score [ Time Frame: immediately after IUD insertion ] | immediately after IUD insertion
  The visual analog scale (VAS ) pain score reported by participants immediately after IUD insertion .Pain scores will be measured using a visual analogue scale (VAS) consisting of a 10 cm horizontal straight line on which 0 cm corresponds to no pain and 10 cm to the worst pain. VAS is rated as 0 for no pain, 1-3 for mild pain, 4-6 for average pain, and 7-9 for severe pain and 10 for extremely severe pain an individual can experience .
  A research assistant standing beside the woman will hold the VAS sheet for the participant to select the point that corresponds to the level of pain she will experience after IUD insertion .

SECONDARY OUTCOMES:
Immediate complications related to IUD insertion [ Time Frame: one day after insertion]: | one day after insertion
  Immediate complications related to IUD insertion [ Time Frame: one day after insertion]:
  The immediate complications related to IUD insertion such as :
  1. Failure of insertion .
  2. Vasovagal reaction .
  3. The number of women who will need analgesics after insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Alhassan M Khedr, Study Director — Ain Shams University
Locations (1):
- AinSHAMS UNIV, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aksoy H, Aksoy U, Ozyurt S, Acmaz G, Babayigit M. Lidocaine 10% spray to the cervix reduces pain during intrauterine device insertion: a double-blind randomised controlled trial. J Fam Plann Reprod Health Care. 2016 Apr;42(2):83-7. doi: 10.1136/jfprhc-2014-100917. Epub 2015 Mar 10. PMID 25759418